CLINICAL TRIAL: NCT03979391
Title: Detecting Oligoclonal Bands Through Isoelectric Focusing of Tears in Children With Radiologically Isolated Syndrome or Clinically Isolated Syndrome: a Diagnostic, Prospective, Multicentric Study With a 2-year Longitudinal Follow-up
Brief Title: Isoelectric Focusing of Tears in Children With Radiologically Isolated or Clinically Isolated Syndrome
Acronym: OBIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0070
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Clinically Isolated Syndrome; Radiologically Isolated Syndrome; Multiple Sclerosis in Children
Keywords: Clinically Isolated Syndrome; Radiologically Isolated Syndrome; Multiple Sclerosis; Children; Tear analysis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with CIS or RIS (Experimental): The detection of supernumerary oligoclonal bands (OCBs) in tears will be performed
  Interventions: Diagnostic Test: Tear collection and lumbar punction

INTERVENTIONS:
Diagnostic Test: Tear collection and lumbar punction — Tear collection and lumbar punction will be performed in order to detect supernumerary oligoclonal bands

SUMMARY:
The main gold of this study is to lead a multicentric, prospective study, to evaluate the diagnostic quality of tears in children with clinically isolated syndrome (CIS) and radiologically isolated syndrome (RIS) during a longitudinal follow-up.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a disease that affects the white matter of the central nervous system. In France, approximately 100,000 patients are affected. It is one of the most common neurological condition in young adults.

The presence of supernumerary oligoclonal bands (OCBs) in the cerebrospinal fluid (CSF) in comparison to the serum was established in 2017 as a criterion for temporal dissemination in MS patients. This is a predictive factor of conversion to MS in the clinically isolated syndrome (CIS) and radiologically isolated syndrome (RIS), either in children or adults.

However, the main inconvenient of OCB analysis in CSF is the requirement of a lumbar puncture, which is a traumatising technique that may raise ethical concerns especially when it has to be performed in children.

Searching for OCBs in tears, which are more accessible, may represent an attractive alternative. Some published articles studying adult populations go in this direction, but there are no data in the literature regarding children.

The main gold of this study is to lead a multicentric, prospective study, to evaluate the diagnostic quality of tears in children with clinically isolated syndrome (CIS) and radiologically isolated syndrome (RIS) during a longitudinal follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age < 18 years old
* informed consent from the child and the parents (at least one of the two legal guardians)
* child covered by social security

For the RIS population:

* asymptomatic child
* fortuitous discovery of lesions strongly suggesting sclerosis multiple on a Magnetic resonance imaging (MRI) scan

For the CIS population:

- child presenting a CIS in the past three months

Exclusion Criteria:

* patient with remitting MS
* patient with progressive MS
* patient with eye infection
* patient under immunosuppressive therapy on the day of inclusion due to the treatment of another disease than MS

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2024-11-26 (Estimated); Study Completion 2024-11-26 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of tears analysis compared to lumbar punction analysis for the diagnosis of CIS and RIS | Day 0
  To evaluate the diagnostic performance of tears analysis in children with CIS and RIS, (sensitivity, specificity, positive and negative predictive value) being the gold standard the cerebrospinal analysis
Specificity of tears analysis compared to lumbar punction analysis for the diagnosis of CIS and RIS | Day 0
  To evaluate the diagnostic performance of tears analysis in children with CIS and RIS, (sensitivity, specificity, positive and negative predictive value) being the gold standard the cerebrospinal analysis
Positive predictive value of tears analysis compared to lumbar punction analysis for the diagnosis of CIS and RIS | Day 0
  To evaluate the diagnostic performance of tears analysis in children with CIS and RIS, (sensitivity, specificity, positive and negative predictive value) being the gold standard the cerebrospinal analysis
Negative predictive value of tears analysis compared to lumbar punction analysis for the diagnosis of CIS and RIS | Day 0
  To evaluate the diagnostic performance of tears analysis in children with CIS and RIS, (sensitivity, specificity, positive and negative predictive value) being the gold standard the cerebrospinal analysis

SECONDARY OUTCOMES:
Proportion of patients with OCBs in tears | day 0, one year

CONTACTS AND LOCATIONS:
Overall Officials: Hautecoeur Patrick, Principal Investigator — Lille Catholic University
Locations (1):
- GHICL, Lomme, France

IPD SHARING:
Plan to Share IPD: No